CLINICAL TRIAL: NCT04159597
Title: Expanded Access to Upadacitinib
Status: Available | Type: Expanded Access
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: C20-082; C25-267 (Other: Abbvie)
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease; Ulcerative Colitis; Idiopathic Arthritis (Including sJIA, pJIA, or JPsA); Atopic Dermatitis
Keywords: Expanded Access; Pre-approval Access; Compassionate Use; Special Access Program; Named Patient Basis; Special Access Scheme
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Dermatitis, Atopic | interventions — upadacitinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Upadacitinib — Upadacitinib will be administered as oral solution.
  Other Names: ABT-494; Rinvoq; C25-267

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to upadacitinib prior to approval by the local regulatory agency. Availability will depend on territory eligibility. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

ELIGIBILITY:
Exclusion Criteria:

* There are other suitable treatment options.
* The participant qualifies for ongoing clinical trials.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie